CLINICAL TRIAL: NCT06593613
Title: Pilot Randomized Trial of the RUBI Program for Families of Autistic Adults
Brief Title: Pilot Trial of the RUBI Program for Autistic Adults
Acronym: RUBI-A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Els for Autism (Unknown); Drexel University (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCH STUDY00004782
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder; Behavior; Parenting
MeSH Terms: conditions — Autism Spectrum Disorder; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RUBI-A (Experimental): Recently redesigned version of the RUBI program for autistic adults and their caregivers
  Interventions: Behavioral: RUBI-A
- R-ISLEA (Active Comparator): Psychoeducation control condition
  Interventions: Behavioral: R-ISLEA

INTERVENTIONS:
Behavioral: RUBI-A — The RUBI-A intervention includes 9 sessions covering Behavioral Principles, Prevention Strategies, Visual Supports, Reinforcement, Co-Regulation, Supporting Communication, Effective Instructions, Teaching Skills, and Generalization and Maintenance. RUBI teaches skills to help build a behavioral "toolbox" for challenging behaviors and adaptive skills. RUBI emphasizes: 1) tailoring the intervention to the specific individual; 2) identifying behavioral function instead of topography to inform behavioral strategy choice; 3) increasing appropriate behaviors; and 4) using positive behavioral supports,39,40 such as antecedent management (e.g., use of visual supports), reinforcement, and functional communication strategies to support independence, self-help, and safety skills.
  Arms: RUBI-A
Behavioral: R-ISLEA — R-ISLEA training focuses on increasing core knowledge and understanding of autism, but it does not provide specific guidance on behavioral strategies for managing challenging behaviors. Developed by autism experts at Drexel University in collaboration with autistic self-advocates, ISLEA is a commercially available psychoeducation program designed for educators, direct support staff, families, caregivers, and autistic individuals. If English is not the language of care for a dyad, subtitles in the preferred language will be provided for the webinars, and interpreters will be available for the live sessions.
  Arms: R-ISLEA

SUMMARY:
The goal of this clinical trial is to evaluate if a redesigned version of the RUBI parenting intervention can reduce challenging behaviors and improve adaptive skills in autistic adults with co-occurring challenging behaviors. The main questions it aims to answer are:

* Is the redesigned RUBI intervention feasible and acceptable for autistic adults and their families?
* Does the redesigned RUBI intervention reduce challenging behaviors and enhance the quality of life for autistic adults?
* Researchers will compare the redesigned RUBI intervention to an active control group, Introduction to the Science and Lived Experience of Autism (ISLEA), to see if RUBI is more effective in improving outcomes for autistic adults and their families.

Participants will:

* Attend sessions where they receive either the RUBI intervention or the ISLEA program.
* Engage in activities designed to promote communication, co-regulation, and autonomy in the context of supporting autistic adults.
* Complete assessments at the start, throughout, and at the end of the 20-week trial to evaluate outcomes such as challenging behaviors, adaptive skills, and quality of life.

DETAILED DESCRIPTION:
Over the past decade, across three large-scale, NIH-funded trials, the Research Unit in Behavioral Interventions (RUBI) Autism Network developed and systematically tested a low-intensity manualized parenting intervention for autistic children ages 3-14 with challenging behaviors.8-10 RUBI teaches families how to foster home environments that support their autistic child, including teaching parents how to understand their child's behaviors as forms of communication, respond and adapt to their child's unique needs, and personalize strategies for their child's needs and preferences (e.g. utilizing visual supports to align with information processing needs; attuning to the negative impact of unpredictable expectations; accommodating sensory needs). RUBI also may be a promising approach to support families as they provide care and support to their autistic adult dependents.

RUBI has been found to be acceptable to families, reliably delivered by trained therapists, and effective in reducing challenging behaviors and increasing adaptive skills in children.8-10 In response to the shortage of efficacious interventions for autistic adults, RUBI could serve to be systematically redesigned to better support collaboration between family members and their autistic adult dependents, thereby helping autistic adults lead more meaningful and independent lives. To this end, RUBI was recently redesigned utilizing the Discover, Design/Build, Test (DDBT) Framework,11 which leverages user-centered design, participatory action research, and implementation science to ensure that a modified intervention meets the needs of end users (parents, autistic adults, community providers) and is viable across contexts (home, community). Redesign targets included (1) changes in text examples, in-session activities, and language to be more acceptable and relevant to the autistic adult population, (2) content modifications to align focus on supporting communication and dyad co-regulation, (3) improvement in inclusionary and collaborative engagement strategies, and (4) promotion of the autistic adult's engagement, autonomy, and agency during sessions and when implementing strategies.

With the Discover, Design/Build phases successfully completed, a two-year pilot randomized trial will extend our work to the Test phase in order to evaluate the feasibility, acceptability, and efficacy of the newly redesigned RUBI intervention compared to an active control - Introduction to the Science and Lived Experience of Autism (ISLEA). Eighty autistic adults with co-occurring challenging behaviors and their parents will be randomized 1:1 to either RUBI or ISLEA and followed for 20 weeks in order to evaluate key outcomes, including feasibility and acceptability of the redesigned RUBI intervention. This study will also explore the impact of RUBI on autistic adults' challenging behaviors, adaptive skills, and quality of life as well as parent self-efficacy. Successful completion of this proposed pilot study will allow for a future large-scale effectiveness trial of RUBI with autistic adults and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Autistic adults will:

  1. be age ≥ 18 years;
  2. live at home with their parent and be able to attend each session;
  3. have a community diagnosis of autism (confirmed through record documentation) and Social Communication Questionnaire (SCQ) total score > 15;
  4. have a parent rated 24-item EDI Reactivity Score > 50 percentile, which reflects mild to moderate challenging behaviors (e.g., outbursts; verbal aggression);
  5. have receptive language > 18 months as measured on the Mullen Scales of Early Learning (MSEL) Receptive Language subtest or similar measure of receptive language;
  6. have a stable educational/vocational plan and be medication free or on stable medication (no changes in prior 6 weeks or planned changes for 16 weeks). Individuals on stable medication will be included as this enhances sample representativeness.
* Parents/Legally Authorized Representatives will be able to:

  1. attend each session.

Exclusion Criteria:

* Autistic adults with: (1) serious medical conditions requiring immediate care (e.g., uncontrolled seizures) or (2) serious behavioral challenges where safety to self and/or others is of concern and that warrant more immediate or intensive treatment (e.g., self-injurious behaviors or aggression resulting in tissue damage). This will be evaluated through case panel with study site Principal Investigators.
* Parents/Legally Authorized Representatives where they are unable to attend weekly virtual or in person sessions over the course of 20 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Emotion Dysregulation Inventory (EDI) | We will use the 24-item Caregiver Reactivity scale for screening, the full 30-item Caregiver form at Baseline, Week 8, Week 16, and Week 20, and the 13-item Self-Report scale at Baseline, Week 8, Week 16, and Week 20.
  The EDI is an informant report measure of emotion dysregulation over the past 7 days, rated on a five-point scale from "not at all" to "very severe." The EDI produces scores for Reactivity and Dysphoria. Cronbach's alpha ranges from .90-.97.
Open Source Challenging Behavior Scale (OS-CBS) | We will administer the OS-CBS to the caregiver at Baseline, Week 8, Week 16, and Week 20.
  The OS-CBS is an 18-item questionnaire that asks caregivers to rate, over the past month, how much of a problem a specific behavior is, using a 5-point Likert Scale (1 = Not at all a problem, 2 = Mild Problem, 3 = Moderate Problem, 4 = Severe Problem, 5 = Very Severe Problem).
Aberrant Behavior Checklist (ABC) | We will administer the ABC to the caregiver at Baseline and Week 20.
  The ABC measures behavioral challenges in individuals with developmental disabilities. It contains 58 items, with 5 subscales: Irritability, Social Withdrawal, Stereotypic Behavior, Hyperactivity/Noncompliance, and Inappropriate Speech. Items are scored from 0 (never a problem) to 3 (severe problem). Higher scores indicate greater problems in that area. The ABC has high subscale internal consistency (mean alpha = 0.91), excellent test-retest reliability (mean r = 0.98), acceptable inter-rater reliability (mean r = 0.63). The ABC has been used in previous RUBI trials and is sensitive to change with intervention.
Home Situations Questionnaire - Autism Spectrum Disorder (HSQ-ASD) | We will administer the HSQ-ASD to the caregiver at Baseline, Week 8, Week 16, and Week 20.
  The HSQ-ASD is a 24-item parent-rated measure of challenging daily routines for autistic individuals. The scale yields per-item mean scores of 0 to 9 (higher scores = greater situational challenges). Based on prior studies, a 25% decrease reflects meaningful improvement in behaviors during daily routine activities.
Top Problems Assessment (TPA) | We will administer the TPA to the caregiver and autistic adult at Baseline and weekly through Week 20.
  The TPA entails gathering severity ratings (scale of 0-4) of the top three problems the autistic adult and parent independently identify as most important to them. Psychometric analyses of the TPA have showed substantial evidence of test-retest reliability (.69-.91), convergent and discriminant validity, and sensitivity to clinical change with treatment.

SECONDARY OUTCOMES:
Adaptive Behavior Assessment System - Third Edition (ABAS-3) | We will administer the ABAS-3 to the caregiver at Baseline and Week 20.
  The ABAS-3 is a norm-referenced measure that assesses adaptive behavior and related skills for individuals from birth through 89 years. Information may be provided by parents or the individual themselves. Scores help describe a person's general adaptive behavior, as well as functioning in 11 related skill areas: Communication, Community Use, Functional Academics, School/Home Living, Health and Safety, Leisure, Self-Care, Self-Direction, Social, Work (for older adolescents and adults), and Motor.
World Health Organization QOL Assessment-Brief (WHO-QOL-BRIEF) | We will administer the WHO-QOL-BRIEF to the autistic adult at Baseline and Week 20.
  The WHO-QOL-BRIEF is a 26-item self-report QoL measure using a 5-point scale, with higher scores indicating better QoL. Questions assess QoL in the domains of physical/psychological health, social relationships, and environment. The WHO-QOL is sensitive to intervention change and has strong internal consistency (α = 0.71-0.82) with autistic adults, who have been shown to accurately report their own QoL (ratings comparable to parents). We will be utilizing both the WHO-QOL-BRIEF, which includes the Disabilities Supplement and Autism Spectrum QoL Supplement.
RUBI Knowledge Assessment and ISLEA Proximal Knowledge Measure | We will administer the knowledge questionnaire to the caregiver and autistic adult at Baseline and Week 16.
  The RUBI Knowledge Assessment and ISLEA Proximal Knowledge Measure were designed by study team members to evaluate intervention-specific knowledge gained from pre to post treatment.
Autism-Specific Parenting Self-Efficacy Scale | We will administer the self-efficacy scale to the caregiver at Baseline and Week 16.
  The Autism-Specific Parenting Self-Efficacy Scale is a 17-item measure of parents' confidence in their ability to manage the unique parenting challenges of raising an autistic child. (mean alpha = 0.91, indicating a high level of internal consistency across scale items).
Zarit-Burden Questionnaire | We will administer the Zarit-Burden scale to the caregiver at Baseline and Week 16.
  The Zarit-Burden Questionnaire is a 22-item measure that reflects how caregivers feel when taking care of another person.
Personal Advocacy Activity Scale (PAAS) | We will administer the PAAS to the autistic adult at Baseline and Week 16.
  The PAAS measures self-reported personal advocacy activities. The PAAS reflects self-reported personal advocacy activities engaged in over the past 3 months. A total of 25 items (e.g., "In the past 3 months, how many times have you arrived organized and prepared for a meeting?") were written using a scale indicating how frequently respondents have engaged in the behavior in the past 3 months (choices were Not at all, 1-2 times, 3- 4 times, and 5 or more times).
New General Self-Efficacy Scale (NGSE) | We will administer the NGSE to the autistic adult at Baseline and Week 16.
  The NGSE is an 8-item measure that assesses how much people believe they can achieve their goals, despite difficulties. Using a 5-point rating scale (1= strongly disagree; 3 = neither agree nor disagree; 5 = strongly agree), respondents show how much they agree with eight statements, such as "Even when things are tough, I can perform quite well." Total scores are calculated by taking the average of all questions.
Rosenberg Self-Esteem Scale (RSES) | We will administer the RSES to the autistic adult at Baseline and Week 16.
  The RSES is a 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self. The scale is believed to be uni-dimensional. All items are answered using a 4-point Likert scale format ranging from strongly agree to strongly disagree.
Autism and Neurodiversity Attitudes Scale (ANAS) | We will administer the ANAS to the autistic adult at Baseline and Week 16.
  The ANAS is a 17-item scale that assesses endorsements of neurodiversity beliefs with respect to autism. The ANAS also contains three subscales - Autism Anti-Stigma, Autism Permanence, and Autism as Difference. All items are answered using a 5-point Likert scale format ranging from strongly disagree to strongly agree.
Neurodiversity Support Scale | We will administer the Neurodiversity - Movement Support to the autistic adult at Baseline and Week 16.
  The Neurodiversity Support Scale is a 8-item scale that assesses how strongly an individual supports the neurodiversity movement. It is adapted from Nario-Redmond et al., 2013. All items are answered using a 7-point Likert scale format ranging from strongly disagree to strongly agree with higher average scores indicting stronger support of the neurodiversity movement.

CONTACTS AND LOCATIONS:
Overall Officials: Daina M Tagavi, PhD, Principal Investigator — Seattle Children's Hospital
Locations (3):
- United States (3):
  - Els for Autism Foundation, Jupiter, Florida
  - A.J. Drexel Autism Institute, Philadelphia, Pennsylvania
  - Seattle Children's Autism Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No